CLINICAL TRIAL: NCT06712901
Title: Social Media and Cancer Screening Information
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Cancer Institute (NCI) (NIH); AmeriSpeak - NORC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HCI183491; 5R37CA259156-04 (NIH)
Record Dates: First submitted 2024-11-19; First posted 2024-12-02 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control (no exposure) (Placebo Comparator): Participants in the Control Arm will not be shown any messages.
  Interventions: Behavioral: Control
- Median Ranked (Experimental): Participants in the Median Ranked Arm will be shown four Median Ranked messages.
  Interventions: Behavioral: Median Ranked Cancer Screening Messaging
- Overall Preferred (Experimental): Participants in the Overall Preferred arm will be shown four Overall Preferred messages.
  Interventions: Behavioral: Overall Preferred Cancer Screening Messaging
- Black American Preferred (Experimental): Participants in the Black American Preferred arm will be shown four Black American Preferred messages.
  Interventions: Behavioral: Black American Preferred Cancer Screening Messaging
- White American Preferred (Experimental): Participants in the White American Preferred arm will be shown four White American Preferred messages.
  Interventions: Behavioral: White American Preferred Cancer Screening Messaging

INTERVENTIONS:
Behavioral: Median Ranked Cancer Screening Messaging — Strong message content that increases screening and sharing intentions. Messages in this intervention were median ranked in the prior study.
  Arms: Median Ranked
Behavioral: Overall Preferred Cancer Screening Messaging — Strong message content that increases screening and sharing intentions. Messages in this intervention were highly rated messages by all participants in the prior study.
  Arms: Overall Preferred
Behavioral: Black American Preferred Cancer Screening Messaging — Strong message content that increases screening and sharing intentions. Messages in this intervention were highly rated messages by Black participants but not White participants in the prior study.
  Arms: Black American Preferred
Behavioral: White American Preferred Cancer Screening Messaging — Strong message content that increases screening and sharing intentions. Messages in this intervention were highly rated messages by White participants but not Black participants.
  Arms: White American Preferred
Behavioral: Control — There will be no message content of cancer screening and sharing intentions in this arm.
  Arms: Control (no exposure)

SUMMARY:
NORC/AmeriSpeak will recruit participants who meet the study criteria and invite them to complete a 15-minute survey. Participants will be randomly assigned to one of five conditions, with approximately 400 people in each condition, and will respond to various questions after viewing the study messaging. Once 2,000 participants complete the survey, the data will be de-identified and provided to the study team for analysis.

DETAILED DESCRIPTION:
NORC/AmeriSpeak will put all of the study content into their system. They will send out the opportunity to participate in the study, which should take about 15 minutes, to people in their panel who meet our participation criteria. Participants will be directed to the study information sheet that includes all elements of consent. Participants who agree to participate will start the survey experiment. The survey experiment will randomize participants into one of five conditions: (1) control (no exposure), (2) overall median ranked messages (from the prior study), (3) messages preferred by all participants, (4) messages preferred by Black American participants, and (5) messages preferred by White American participants. Approximately 400 people will complete each condition. After viewing the study stimuli (or no stimuli in the control condition), participants will respond to various outcomes and other variables of interest (see questionnaire draft included). After all 2,000 people have completed the study, the study team will receive a de-identified data file from NORC/AmeriSpeak with all study data and engage in analysis. This study is planned to close the study around that time as the study team completes data analysis and write-up the findings.

ELIGIBILITY:
Inclusion Criteria:

* Identify as white/Caucasian or Black/African American.

Exclusion Criteria:

* Do not identify as white/Caucasian or Black/African American.
* Previously diagnosed with colorectal cancer
* Non-English speakers

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2030 (Actual)
Dates: Start 2025-01-09 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-01-21 (Actual)

PRIMARY OUTCOMES:
Intentions to adhere to colorectal cancer screening (CRCS) recommendations | 15 minutes
  After reading cancer screening (CRCS) recommendations, this outcome will assess how likely they are to follow on the the screening recommendations.
  Response options: Very unlikely (1), unlikely, neither unlikely nor likely, likely, very likely (5)
  A higher score indicates a favorable outcome, and a lower score indicates a less favorable outcome.
Intentions to adhere test preference indication | 15 minutes
  To determine which colorectal cancer screening (CRCS) participants are most likely to choose.
  Response options: stool-based tests (e.g., FOBT or FIT); endoscopic/scoping approach (e.g., colonoscopy or sigmoidoscopy); whatever my doctor recommends to me; something other than a stool-based or scoping approach; I would not follow the recommendations.
  This outcome will report the count of responses.

SECONDARY OUTCOMES:
Likelihood of sharing information via social media | 15 minutes
  This outcome measure will determine how likely participants are to share the messages about colon cancer screening on social media.
  Response options: Very unlikely (1), unlikely, neither unlikely nor likely, likely, very likely (5)
  A higher score indicates a favorable outcome, and a lower score indicates a less favorable outcome.
Information sharing behavior | 15 minutes
  This outcome will determine the proportion of participants will seek more information after the study.
  The participants will be asked a question on if they would like more information (Yes/No) and survey vendor will track participants who click a link to an external resource like the American Cancer Society to learn more.

CONTACTS AND LOCATIONS:
Overall Officials: Andy King, PhD, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (1):
- Andy King, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared/uploaded to an online data repository like OSF.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Once the primary results are published in a peer-reviewed journal article, the de-identified data will be published in an online data repository. The data will then be available for as long as the online repository is available